CLINICAL TRIAL: NCT06625073
Title: Randomized Trial of Sodium-glucose Cotransporter 2 Inhibition in Heart Transplant Recipients
Brief Title: Randomized Trial of SGLT2i in Heart Transplant Recipients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEPH-004-24S
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplant; Cardiovascular Disease; Kidney Disease
Keywords: Heart Transplant; Empagliflozin; Safety and Tolerability; Kidney Outcomes; Cardiometabolic Outcomes; Erythropoiesis; Functional Status; Quality of Life
MeSH Terms: conditions — Cardiovascular Diseases; Kidney Diseases | interventions — empagliflozin; Control Groups

STUDY DESIGN:
Intervention Model Description: Empagliflozin 10 ng daily for 12 months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects will be randomized to either empagliflozin 10 mg daily for 12 months or matching placebo. The subjects and the investigators will not know whether subjects are randomized to active arm (empagliflozin) or to control arm (placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental): A starting dose of empagliflozin 10 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Participating subjects will remain at this dose for the whole study duration of 12 months.
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): A starting dose of empagliflozin 10 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Participating subjects will remain at this dose for the whole study duration of 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — A starting dose of empagliflozin 10 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Participating subjects will remain at this dose for the whole study duration of 12 months.
  Other Names: Jardiance
  Arms: Empagliflozin
Drug: Placebo — A starting dose of empagliflozin 10 mg or matching placebo will be initiated after randomization and completion of the baseline testing. Participating subjects will remain at this dose for the whole study duration of 12 months.
  Other Names: Control Group
  Arms: Placebo

SUMMARY:
Heart transplant (HTx) is an established therapy for advanced heart disease that restores quality of life and improves survival. However, due to preexisting comorbidities combined with the immunosuppressive therapies required after transplantation, HTx recipients remain at high risk for kidney, cardiovascular (CV), and metabolic disease. Large randomized clinical trials have recently shown that sodium-glucose cotransporter 2 inhibitors (SGLT2i) have potent kidney protective and CV benefits in many populations of patients with chronic kidney disease (CKD), CV disease and/or diabetes. SGLT2i have not been studied prospectively in HTx recipients, which represents a barrier to their use in this population.

In this multicenter randomized controlled trial in Veterans with HTx, investigators will evaluate the potential benefits of empagliflozin on kidney function, cardiometabolic risk, erythropoiesis, and functional status. A total of 200 Veterans will be randomly assigned to receive either empagliflozin 10 mg daily or a matching placebo for 12 months.

DETAILED DESCRIPTION:
Heart transplant (HTx) markedly improves patient health-related quality of life (hrQoL) and survival in advanced heart failure (HF). However, HTx recipients remain at elevated risk for kidney and cardiovascular (CV) morbidity and mortality. Mitigating the negative effects of these morbidities on long-term survival and on patient hrQoL after HTx is a critical unmet need. Large clinical trials have recently shown that sodium glucose cotransporter 2 inhibitors (SGLT2i) have potent kidney protective and CV benefits. By preventing glucose reabsorption in the renal proximal tubule and promoting glycosuria, SGLT2i trigger multiple downstream effects, including improvement in insulin sensitivity and in mitochondrial efficiency in kidney and heart. SGLT2i also modulate sympathetic activity, improve endothelial function and reduce inflammation, with resultant improvement in myocardial and vascular function. SGLT2i increase erythropoietin levels and improve iron utilization. HTx is often complicated by development of chronic kidney disease (CKD), diabetes mellitus (T2D), anemia, and CV events, especially cardiac allograft vasculopathy (CAV). Although SGLT2i may significantly reduce development of these complications, prospective studies of SGLT2i did not include transplant recipients, leaving an important knowledge gap. HTx recipients could derive particularly significant benefits from SGLT2i therapy. The investigators hypothesize that SGLT2i with empagliflozin in HTx recipients will result in beneficial effects on kidney function, cardiometabolic risk, erythropoiesis and functional status, and that SGLT2i use in this population will be safe and well tolerated. The specific aims of this study are:

Specific Aim 1. Investigate the effects of SGLT2i with empagliflozin on kidney function in HTx recipients.

Kidney disease after HTx is a potent predictor of mortality. Investigators hypothesize that treatment with empagliflozin will preserve kidney function after HTx.

Aim 1a. Assess the effects of SGLT2i on urinary albumin-to-creatinine ratio (UACR). Albuminuria, represented by UACR and an independent predictor of kidney outcomes, was consistently reduced by SGLT2i in the landmark trials of SGLT2i. Approximately 50% of Veterans after HTx have at least moderate albuminuria. Investigators hypothesize that empagliflozin therapy will decrease albuminuria in HTx recipients.

Aim 1b. Assess the effect of SGLT2i on estimated glomerular filtration rate (eGFR).

SGLT2i therapy was associated with significantly slower decline of eGFR in all SGLT2i clinical trials of CKD. Investigators hypothesize that empagliflozin treatment will result in an improvement of eGFR slope in HTx recipients.

Specific Aim 2. Establish the safety and tolerability of SGLT2i therapy in HTx recipients.

SGLT2i have been tested prospectively in >75,000 patients and demonstrated a favorable safety profile. Exclusion of organ transplant recipients from these trials resulted in an important knowledge gap-the lack of safety and tolerability data in this population, which limits clinicians' use of SGLT2i in HTx recipients. Investigators hypothesize that treatment with empagliflozin in HTx recipients will be associated with favorable safety and tolerability.

Specific Aim 3. Evaluate the cardiometabolic, erythropoietic and functional effects of SGLT2i after HTx.

Cardiometabolic risks in HTx recipients contribute to CAV, graft failure, functional limitations and mortality. Investigators hypothesize that empagliflozin therapy will result in favorable cardiometabolic, erythropoietic and functional effects.

Aim 3a. Assess the effects of SGLT2i on markers of cardiometabolic risk.

Investigators will examine the effect of empagliflozin on hemoglobin A1c (HbA1c), body weight and blood pressure (BP), inflammation and on cardiac allograft health assessed through cardiac imaging and cardiac biomarkers. Investigators hypothesize that empagliflozin therapy will result in favorable cardiometabolic effects.

Aim 3b. Assess the effects of SGLT2i on erythropoiesis.

SGLT2i stimulates erythropoiesis, but the exact mechanisms are not well understood. Investigators hypothesize that empagliflozin will result in an increase in serum erythropoietin and amelioration of anemia in HTx recipients.

Aim 3c. Assess the effects of SGLT2i on functional status and health-related quality of life.

SGLT2i have improved functional status and hrQoL in non-transplant populations. Investigators hypothesize that the favorable kidney, cardiometabolic and erythropoietic effects of empagliflozin after HTx will result in a corresponding increase in six-minute walk test (6MWT) and hrQoL after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Heart transplant recipient, 3 months after transplant

Exclusion Criteria:

1. eGFR <20 mL/min/1.73m2
2. Type 1 diabetes mellitus
3. HbA1C >10%
4. Baseline UACR <30 mg/g in patients without T2D
5. Known allergy or intolerance to SGLT2i
6. Active uncontrolled infection
7. Multiorgan transplant
8. SGLT2i treatment in the last 30 days
9. Pregnancy, breast-feeding or woman of child-bearing age not on birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin-to-creatinine ratio (UACR) | 12 months
  UACR difference (mg/g) in subjects in active arm vs control arm
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12 months
  Adverse and serious adverse events difference in active arm vs control arm

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate (eGFR) | 12 months
  eGFR difference (mL/min/1.73m2) in subjects in active arm vs control arm
Hemoglobin A1c (HbA1c) | 12 months
  HbA1c difference (%) in subjects in active arm vs control arm
Fasting blood glucose | 12 months
  Fasting blood glucose difference (mg/dL) in subjects in active arm vs control arm
Body weight | 12 months
  Body weight difference (kg) in subjects in active arm vs control arm
Systolic and diastolic blood pressure | 12 months
  Systolic and diastolic blood pressure difference (mmHg) in subjects in active arm vs control arm
Serum high sensitivity C-reactive protein (hsCRP) | 12 months
  Serum hsCRP difference (mg/L) in subjects in active arm vs control arm
Serum N-Terminal Pro-B-Type Natriuretic Peptide (NTproBNP) | 12 months
  Serum NTproBNP difference (pg/mL) in subjects in active arm vs control arm
Hemoglobin | 12 months
  Hemoglobin difference (g/dl) in subjects in active arm vs control arm
Serum erythropoietin | 12 months
  Serum erythropoietin difference (mU/mL) in active arm vs control arm
Hematocrit | 12 months
  Hematocrit difference (%) in active arm vs control arm
Serum transferrin saturation | 12 months
  Serum transferrin saturation difference (%) in active arm vs control arm
Six Minute Walk Test | 12 months
  Difference in distance (m) covered in the 6 minute walk test in active arm vs control arm
Serum high sensitivity Troponin | 12 months
  Serum high sensitivity Troponin difference (pg/mL) in subjects in active arm vs control arm
Kansas City Cardiomyopathy Questionnaire-12 | 12 months
  Kansas City Cardiomyopathy Questionnaire-12 overall summary score difference in active arm vs control arm. Scale range 0-100. Higher result is better.
Serum tumor necrosis factor -a (TNF-a) | 12 months
  TNF-a difference (pg/mL) in subjects in active arm vs control arm
Serum interleukin 6 (IL-6) | 12 months
  IL-6 difference (pg/mL) in subjects in active arm vs control arm
Serum interleukin 1b(IL-1b) | 12 months
  IL-1b difference (pg/mL) in subjects in active arm vs control arm

CONTACTS AND LOCATIONS:
Overall Officials: Josef Stehlik, MD MPH, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (6):
- United States (6):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No